CLINICAL TRIAL: NCT03076541
Title: Cardiovascular Variability, Heart Rate Response, and Electromyogram Power Associated With Periodic Leg Movements.
Acronym: PLMS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1700175
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome; Periodic leg movements; Heart rate; Heart rate variability; Microarousals; Autonomic nervous system activity
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with restless legs syndrome
  Interventions: Device: standard 24-h ambulatory polysomnography

INTERVENTIONS:
Device: standard 24-h ambulatory polysomnography — A standard 24-h ambulatory ad libitum polysomnography including EEG, electro-oculography (EOG), electromyography (EMG), EKG, was performed by a standard clinical.

SUMMARY:
Periodic leg movements during sleep is associated with microarousals and a stimulation of the sympathetic nervous system. The knowledge of this autonomic activation may help understanding the increase of cardiac risk observed in elderly. The aim of the study is to evaluate the relationship between periodic leg movements severity, age, gender, electromyographic power and heart rate response associated with periodic leg movements. Drug-free patients diagnosed with periodic leg movements were included. Clinical data and 24-h polysomnography recordings were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Restless legs syndrome patients
* Hospital routine for periodic leg movements diagnosis
* PLMS index > 0

Exclusion Criteria:

* Narcolepsy-cataplexy
* Sleep irregularities and sleep deprivation symptoms
* Lack of neurological or psychiatric diseases
* Upper airway resistance syndrome
* Obstructive sleep apnea
* Treatment, cerebral lesion, medical illness
* Medication or drinks affecting sleep and wake state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with restless legs syndrome with a diagnosis from January 1rst 2012 to september 1rst 2016.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Amplitude of heart rate response associated with periodic leg movements. | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography

SECONDARY OUTCOMES:
Other Heart rate variability indices: Ptot, very-low-frequency (VLF), low frequency (LF), low frequency normalized units (LFnu), high-frequency normalized units (HFnu), LF/HF. | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography
electromyography (EMG) power | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PICHOT, PhD, Study Chair — CHU SAINT-ETIENNE; Emilia SFORZA, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No